CLINICAL TRIAL: NCT00069277
Title: A Phase I Dose-Finding Study of E7389 (Halichondrin B Analog) Administered Once Every Three Weeks in Patients With Advanced Solid Tumors
Brief Title: Study of E7389 Administered Once Every 3 Weeks In Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Dale Shuster, Ph.D, Eisai Medical Research
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7389-A001-102
Record Dates: First submitted 2003-09-19; First posted 2003-09-24 (Estimated); Results first posted 2012-02-09 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Cancer
Keywords: Cancer, tumors
MeSH Terms: conditions — Neoplasms | interventions — eribulin

INTERVENTIONS:
Drug: E7389

SUMMARY:
The malignancies (advanced solid tumors) that have been chosen for evaluation of E7389 are those where E7389 has demonstrated significant pre-clinical anti-tumor activity, both in vitro and in vivo. The ultimate goal is to demonstrate the clinical activity of E7389 in the treatment of these, and potentially other, tumor types.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically or cytologically confirmed and measurable advanced solid tumor that has progressed following standard therapy or for which no standard therapy exists (including surgery or radiation therapy)
* Patients may have received prior chemotherapy (limit of two prior chemotherapy regimens)
* Patients must be aged >= 18 years
* Patients must have a Karnofsky Performance Status of > 70% -- Patients must have a life expectancy of > 3 months
* Patients must have adequate renal function as evidenced by serum creatinine <1.5 mg/dL or creatinine clearance > 60 mL/minute
* Patients must have adequate bone marrow function as evidenced by absolute neutrophil count > 1,500/µL and platelets > 100,000/µL
* Patients must have adequate liver function as evidenced by bilirubin < 1.5 mg/dL and alanine transaminase (ALAT) and aspartate transaminase (ASAT) < 2 times the upper limits of normal
* Patients must be willing and able to comply with the study protocol for the duration of the study
* Patients must give written informed consent prior to any study-specific screening procedures with the understanding that the patient may withdraw consent at any time without prejudice.

Exclusion Criteria:

* Patients who have received chemotherapy within three weeks (six weeks if nitrosoureas were received) of E7389 treatment start
* Patients who have not recovered from any chemotherapy related or other therapy related toxicity at study entry
* Patients who require therapeutic doses of anti-coagulant therapy (eg, Coumadin, heparin, low molecular weight heparin). Low doses of anticoagulants used for patency (e.g., lines, catheters, ports) are permitted.
* Women who are pregnant or breastfeeding.
* Women of childbearing potential with either a positive pregnancy test at Screening or no pregnancy test. Women of childbearing potential unless (1) surgically sterile or (2) using adequate measures of contraception in the opinion of the Investigator (postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential)
* Fertile men who are not willing to use contraception or fertile men with a female partner who is not willing to use contraception
* Patients who have not successfully completed local therapy for previously treated central nervous system (CNS) metastases and who have not been discontinued from corticosteroids for at least four weeks before starting treatment with E7389. Patients with asymptomatic brain metastases who have no evidence of midline shift on CT scan or MRI may be enrolled without initiation of local therapy for the CNS metastases. In this case, a repeat scan must be performed within four weeks of the original scan to ensure that disease progression is not occurring.
* Patients who have tested positive for HIV
* Patients with severe uncontrolled intercurrent illness/infection (excluding malignancies)
* Patients with cardiovascular impairment
* Patients with organ allografts
* Patients who have received investigational drugs, including immunotherapy, gene therapy, hormone therapy, or other biologic therapy; anti-neoplastic therapy; or radiation therapy (other than required for palliation) within three weeks of E7389 treatment start
* Patients who have had major surgery within four weeks of E7389 treatment start without a full recovery
* Patients with a hypersensitivity to Halichondrin B and/or Halichondrin B-like compounds Patients with other significant disease that, in the Investigator's opinion, would exclude the patient from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2003-08; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dale Schuster, Ph.D, Study Director — Eisai Inc.
Locations (3):
- United States (3):
  - Cancer Institute Medical Group, Los Angeles, California
  - Premiere Oncology, Santa Monica, California
  - New Brunswick, New Jersey

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 2 centers in U.S.during the period of Aug 2003 to Apr 2005.
Groups:
- E7389 Dose-Escalating: E7389 dose-escalation starting at 0.25 mg/m^2 intravenous on Day 1 of a 21 day cycle. Dose escalations scheme used a two part design and proceeded based on dose-limiting toxicity and maximum tolerated dose.
Period: Overall Study
Arm/Group | E7389 Dose-Escalating
Started | 21
Completed | 0
Not Completed | 21
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — Progressive Disease | 15
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | E7389 Dose-Escalating
Number analyzed (Participants) | 21
Age, Customized [Mean (Standard Deviation); unit: participants]
  Mean (+/- Standard Deviation) | 59.0 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
  Hispanic/Latino | 3

OUTCOME MEASURES:

1. Primary Outcome: Response and Progression Will be Evaluated in This Study Using the New International Criteria Proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee. Changes in Only the Largest Diameter of the Tumor Lesions Are Used.
Time Frame: 12 Weeks
Measure: Number; unit: participants
Arm/Group | E7389 Dose-Escalating
Number analyzed (Participants) | 21
participants
  partial response | 1
  stable disease | 12
  progressive Disease | 7

ADVERSE EVENTS:
Arm/Group | E7389 Dose-Escalating
Serious Adverse Events (participants affected / at risk) | 10/21
Other Adverse Events (participants affected / at risk) | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E7389 Dose-Escalating (N=21)
Ileus (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
Hyponatremia (Investigations) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 6
Pyrexia (General disorders) | 1
Infection (Infections and infestations) | 1
Headache (Nervous system disorders) | 1
Fatigue (General disorders) | 1
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Bacteremia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Dysphagia (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E7389 Dose-Escalating (N=21)
Anemia (Blood and lymphatic system disorders) | 6
Febrile Neutropenia (Blood and lymphatic system disorders) | 6
Leukopenia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Tachycardia (Cardiac disorders) | 2
Abdominal Distention (Gastrointestinal disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 6
Diarrhea (Gastrointestinal disorders) | 3
Dry Mouth (Gastrointestinal disorders) | 2
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 2
Chest Pain (General disorders) | 3
Fatigue (General disorders) | 11
Mucosal Inflammation (General disorders) | 2
Peripheral Edema (General disorders) | 3
Pyrexia (General disorders) | 3
Oral Candidiasis (Infections and infestations) | 2
Upper Respiratory Tract Infection (Infections and infestations) | 2
Urinary Tract Infection (Infections and infestations) | 2
Alanine Aminotransferase Increased (Investigations) | 3
Blood Alkaline Phosphatase Increased (Investigations) | 2
Weight Decreased (Investigations) | 4
White Blood Cell Count Decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 4
Decreased Appetite (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 5
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 3
Dysuria (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea Exertional (Respiratory, thoracic and mediastinal disorders) | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 7
Dry Skin (Skin and subcutaneous tissue disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Night Sweats (Skin and subcutaneous tissue disorders) | 3
Pruritis (Skin and subcutaneous tissue disorders) | 4
Rash Pruritic (Skin and subcutaneous tissue disorders) | 2
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No